CLINICAL TRIAL: NCT01782651
Title: Treatment Options in Human Epidermal Growth Factor Receptor 2 (HER2) Positive Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116450
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasms, Breast
Keywords: HER2 positive; Breast Cancer; treatment patterns
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HER2+ metastatic breast cancer patients treated with lapatinib: HER2+ metastatic breast cancer patients treated with lapatinib plus capecitabine
  Interventions: Drug: Lapatinib plus capecitabine

INTERVENTIONS:
Drug: Lapatinib plus capecitabine — Lapatinib plus capecitabine

SUMMARY:
This study will describe the treatment paradigm used over recent years in the clinical management of Human Epidermal Growth Factor Receptor 2 (HER2)+ metastatic breast cancer in Hungary. This information will provide insight into real-world exposure and adherence to anti-HER2 therapy containing regimens, and improve understanding of the reasons for discontinuation of this therapy.

This is a retrospective, descriptive, cohort study of approximately 180 female patients diagnosed with HER2-positive metastatic breast cancer in Hungary. Patients diagnosed with, or who progressed to, metastatic disease between 01 September 2009 and 01 September 2010 will be included. All patients will be followed until death, loss to follow-up or the end of the study period (30 September 2012). All data will be collected retrospectively from patient medical records.

Descriptive statistics of the demographic and clinical characteristics of HER2+ metastatic breast cancer patients, including sites of metastases, the time from initial breast cancer diagnosis until diagnosis of metastatic disease, and HER2 testing methodology and status of HER2 will be described. Further, descriptive statistics of the proportion of HER2+ metastatic breast cancer patients who received anti-HER2 therapy, the sequencing of different therapies, and the duration of therapies in the metastatic setting will be analysed. Among the subset of women who receive lapatinib plus capecitabine, descriptive statistics of the timing of initiation of lapatinib plus capecitabine in the metastatic treatment pathway, time to treatment discontinuation and time to progression (TTP) on lapatinib plus capecitabine will be calculated. Further, descriptive statistics of the type and duration anti-HER2 therapies used prior to initiation of lapatinib plus capecitabine and, where relevant, after lapatinib+capecitabine will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older at diagnosis of, or progression to, metastatic breast cancer
* Patients with a diagnosis of breast cancer with documented metastatic disease and with known date of metastatic disease
* Patients with a histologically confirmed HER2+ breast cancer (HER2 testing procedures per routine institutional practice; no tissue re-sampling will be performed. If conducted at another site, documented results must be available).

Exclusion Criteria:

* Patients receiving care for another primary cancer during the study time period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to capture data on approximately 180 patients with HER2-positive metastatic breast cancer in about 20 medical centres in Hungary. Patients diagnosed with, or who progressed to, metastatic disease between 01 September 2009 and 01 September 2010 will be included. All patients will be followed until death, loss to follow-up or the end of the study period (30 September 2012).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) expressed in weeks and months | 2 years

SECONDARY OUTCOMES:
Time to discontinuation of lapatinib plus capecitabine, expressed in weeks and months. | 2 years
  Discontinuation will be measured from the initiation of lapatinib plus capecitabine to the date of discontinuation of this regimen due to any reason. Patients still responding to lapatinib plus capecitabine at the end of the Follow up Period will be censored at the date of the last follow-up contact.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Debrecen, Hungary